CLINICAL TRIAL: NCT00844753
Title: Atomoxetine, Placebo and Parent Management Training in Autism
Acronym: Strattera
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: University of Pittsburgh (Other); Ohio State University (Other)
Responsible Party: Principal Investigator, tristram smith, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R01MH079082-01A2 (NIH); NCT00699205 (obsolete NCT alias)
Record Dates: First submitted 2008-06-06; First posted 2009-02-16 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Autism; Pervasive Development Disorder; Asperger's Disorder; Attention Deficit Hyperactivity Disorder
Keywords: Autism; PDD NOS; Attention Deficit Hyperactivity Disorder; Parent Management Training
MeSH Terms: conditions — Autistic Disorder; Child Development Disorders, Pervasive; Asperger Syndrome; Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Atomoxetine + Parent Management Training
  Interventions: Drug: atomoxetine; Behavioral: Parent Management Training
- 2 (Active Comparator): Atomoxetine without Parent Management Training
  Interventions: Drug: atomoxetine
- 3 (Placebo Comparator): Placebo + Parent Management Training
  Interventions: Drug: Placebo; Behavioral: Parent Management Training
- 4 (Placebo Comparator): Placebo without Parent Management Training
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: atomoxetine — atomoxetine
  Arms: 1; 2
Drug: Placebo — Placebo + parent management treatment
  Arms: 3; 4
Behavioral: Parent Management Training
  Arms: 1; 3

SUMMARY:
The study will evaluate the effectiveness of atomoxetine (Strattera) with and without Parent Management Training (PMT) in children with Autism, Asperger's Disorder, or Pervasive Developmental Disorder Not Otherwise Specified (PDDNOS) who have symptoms of Attention Deficit Hyperactivity Disorder (ADHD). This is a double-blind placebo, parallel study where the atomoxetine will have a dose titration over a 6 week period. All children will be seen weekly during this titration period, with additional visits at Week 8 and Week 10. Families assigned to the PMT arm will have an additional weekly meeting with a clinician for a total of 9 PMT visits. PMT involves teaching parents to implement behavioral interventions with their children. Subjects who are clinical responders (ADHD Responders and Compliance Responders) from the 10 week study period will be followed every 4 weeks in a 24-week extension study. Subjects who are clinical nonresponders will continue in PMT if they received PMT during the double-blind phase, and they will receive an open trial of atomoxetine if they were on placebo during the double-blind phase. All subjects (responders and nonresponders) will be invited to participate in follow-up assessments every 4 weeks for 24 weeks after the completion of the double-blind phase.

ELIGIBILITY:
Inclusion Criteria:

* Children 5 yrs to 14 years 11 mos with clinical diagnosis of Autism, Asperger's Disorder, or PDDNOS based upon the ADI-R and clinical evaluation by DSM-IV criteria,
* Mental age equal to or greater than 24 months,
* ADHD symptoms based upon the CASI and clinical confirmed diagnosis,
* CGIS-S rating of 4 or grater for ADHD symptoms,
* A mean item score of >1.5 on both the Parent and Teacher (non-parent caregiver) SNAP-IV 18 ADHD symptoms or the 9-symptom hyperactive-impulsive subscale (symptoms must be cross-situational),
* Reliable care provider available to bring subject to clinic visits and weekly sessions.

Exclusion Criteria:

* DSM-IV diagnosis of schizophrenia, schizoaffective disorder psychotic disorder NOS,bipolar disorder, or major depression (if accompanied by a family history of bipolar disorder) based upon evidence of suicidality, CASI, and clinical interview/history,
* Prior failed adequate trial of atomoxetine,
* Use of other psychotropic medications that produce CNS effects,
* Diagnosis of bipolar disorder, major depression, hypertension, cardiovascular disease, narrow angle glaucoma, other significant physical illness,
* Pregnancy or sexually active females (intercourse in the past 6 months, reported by either the subject or caregiver),
* Currently on effective medication treatment for ADHD,
* Prior involvement in Parent Management Training or other similar program,
* Currently on albuterol or taking beta blockers,
* Taking supplements or other complementary medical treatments where dose cannot be held at current level for duration of study

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2008-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Handen, PhD, Principal Investigator — University of Pittsburgh Medical Center; Michael Aman, PhD, Principal Investigator — Ohio State University; Tristram Smith, PhD, Principal Investigator — University of Rochester
Locations (3):
- United States (3):
  - University of Rochester Medical Center, Rochester, New York
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Chowdhury M, Aman MG, Scahill L, Swiezy N, Arnold LE, Lecavalier L, Johnson C, Handen B, Stigler K, Bearss K, Sukhodolsky D, McDougle CJ. The Home Situations Questionnaire-PDD version: factor structure and psychometric properties. J Intellect Disabil Res. 2010 Mar;54(3):281-91. doi: 10.1111/j.1365-2788.2010.01259.x. PMID 20377705
- [Result] Barkley, R. A., & Edelbrock, C. (1987). Assessing situational variation in children's problem behaviors: The Home and School Situations Questionnaires. In R. Prinz (Ed.), Advances in behavioral assessment of children and families (pp. 157-176). Greenwich, CT: JAI Press Inc
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] Arnold LE, Ober N, Aman MG, Handen B, Smith T, Pan X, Hyman SL, Hollway J, Lecavalier L, Page K, Rice R Jr. A 1.5-Year Follow-Up of Parent Training and Atomoxetine for Attention-Deficit/Hyperactivity Disorder Symptoms and Noncompliant/Disruptive Behavior in Autism. J Child Adolesc Psychopharmacol. 2018 Jun;28(5):322-330. doi: 10.1089/cap.2017.0134. Epub 2018 Apr 25. PMID 29694241
- [Derived] Lecavalier L, Pan X, Smith T, Handen BL, Arnold LE, Silverman L, Tumuluru RV, Hollway J, Aman MG. Parent Stress in a Randomized Clinical Trial of Atomoxetine and Parent Training for Children with Autism Spectrum Disorder. J Autism Dev Disord. 2018 Apr;48(4):980-987. doi: 10.1007/s10803-017-3345-4. PMID 29022125
- [Derived] Smith T, Aman MG, Arnold LE, Silverman LB, Lecavalier L, Hollway J, Tumuluru R, Hyman SL, Buchan-Page KA, Hellings J, Rice RR Jr, Brown NV, Pan X, Handen BL. Atomoxetine and Parent Training for Children With Autism and Attention-Deficit/Hyperactivity Disorder: A 24-Week Extension Study. J Am Acad Child Adolesc Psychiatry. 2016 Oct;55(10):868-876.e2. doi: 10.1016/j.jaac.2016.06.015. Epub 2016 Aug 2. PMID 27663942
- [Derived] Handen BL, Aman MG, Arnold LE, Hyman SL, Tumuluru RV, Lecavalier L, Corbett-Dick P, Pan X, Hollway JA, Buchan-Page KA, Silverman LB, Brown NV, Rice RR Jr, Hellings J, Mruzek DW, McAuliffe-Bellin S, Hurt EA, Ryan MM, Levato L, Smith T. Atomoxetine, Parent Training, and Their Combination in Children With Autism Spectrum Disorder and Attention-Deficit/Hyperactivity Disorder. J Am Acad Child Adolesc Psychiatry. 2015 Nov;54(11):905-15. doi: 10.1016/j.jaac.2015.08.013. Epub 2015 Sep 3. PMID 26506581

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 200 participants were screened. 131 passed screening. Participants failed screening for the following reasons: 16 Attention Deficit Hyperactivity Disorder (ADHD) not confirmed, 23 Autism Spectrum Disorder not confirmed, 7 previous parent therapy or mental age too low, 23 for other reasons.
Pre-assignment Details: Two participants who passed screening withdrew and one child became ineligible because of ADHD severity declining at baseline.
Groups:
- Atomoxetine (ATX) + Parent Management Training: ATX doses were split twice daily to prevent side effects. However, once-daily dosing was allowed if strongly preferred by a given family. ATX doses were individually adjusted according to a weight-based dosage schedule, with medical clinicians allowed to delay increases or to reduce doses due to adverse events. The initial dose was 0.3 mg/kg/day (rounded to the nearest 5 mg) with weekly escalations by 0.3 mg/kg/day, unless there were limiting side effects or no further room for improvement, to a target dose of 1.2 mg/kg/day, and could be increased to a maximum of 1.8 mg/kg/day based on clinical status and response.
  Parent Management Training (PT)-Families assigned to PT met weekly for individual sessions with a PT clinician. Sessions were adapted from the RUPP Parent Training Manual and covered topics such as preventing behavior problems, reinforcement, time out, and planned ignoring. Each session lasted 60 to 90 minutes and included didactic materials, videos, and role playing.
- Atomoxetine (ATX) Without Parent Management Training: ATX doses were split twice daily to prevent side effects. However, once-daily dosing was allowed if strongly preferred by a given family. ATX doses were individually adjusted according to a weight-based dosage schedule, with medical clinicians allowed to delay increases or to reduce doses due to AEs. The initial dose was 0.3 mg/kg/day (rounded to the nearest 5 mg) with weekly escalations by 0.3 mg/kg/day, unless there were limiting side effects or no further room for improvement, to a target dose of 1.2 mg/kg/day, and could be increased to a maximum of 1.8 mg/kg/day based on clinical status and response.
- Placebo + Parent Management Training: Sugar pill administered twice daily
  Parent Management Training-Families assigned to PT met weekly for individual sessions with a PT clinician. Sessions were adapted from the RUPP Parent Training Manual and covered topics such as preventing behavior problems, reinforcement, time out, and planned ignoring. Each session lasted 60 to 90 minutes and included didactic materials, videos, and role playing.
- Placebo Without Parent Management Training: Sugar pill administered twice daily.
Period: Overall Study
Arm/Group | Atomoxetine (ATX) + Parent Management Training | Atomoxetine (ATX) Without Parent Management Training | Placebo + Parent Management Training | Placebo Without Parent Management Training
Started | 32 | 32 | 32 | 32
Completed | 24 | 29 | 25 | 21
Not Completed | 8 | 3 | 7 | 11
Not completed — Lack of Efficacy | 1 | 0 | 2 | 2
Not completed — Adverse Event | 3 | 2 | 5 | 5
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1
Not completed — could not swallow medication | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Atomoxetine + Parent Management Training: ATX doses were split twice daily to prevent side effects. However, once-daily dosing was allowed if strongly preferred by a given family. ATX doses were individually adjusted according to a weight-based dosage schedule, with medical clinicians allowed to delay increases or to reduce doses due to AEs. The initial dose was 0.3 mg/kg/day (rounded to the nearest 5 mg) with weekly escalations by 0.3 mg/kg/day, unless there were limiting side effects or no further room for improvement, to a target dose of 1.2 mg/kg/day, and could be increased to a maximum of 1.8 mg/kg/day based on clinical status and response.
  Parent Management Training-Families assigned to PT met weekly for individual sessions with a PT clinician. Sessions were adapted from the RUPP Parent Training Manual and covered topics such as preventing behavior problems, reinforcement, time out, and planned ignoring. Each session lasted 60 to 90 minutes and included didactic materials, videos, and role playing.
- Atomoxetine Without Parent Management Training: ATX doses were split twice daily to prevent side effects. However, once-daily dosing was allowed if strongly preferred by a given family. ATX doses were individually adjusted according to a weight-based dosage schedule, with medical clinicians allowed to delay increases or to reduce doses due to AEs. The initial dose was 0.3 mg/kg/day (rounded to the nearest 5 mg) with weekly escalations by 0.3 mg/kg/day, unless there were limiting side effects or no further room for improvement, to a target dose of 1.2 mg/kg/day, and could be increased to a maximum of 1.8 mg/kg/day based on clinical status and response.
- Total: Total of all reporting groups
Arm/Group | Atomoxetine + Parent Management Training | Atomoxetine Without Parent Management Training | Placebo + Parent Management Training | Placebo Without Parent Management Training | Total
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.0 (1.9) | 8.6 (2.3) | 7.7 (1.5) | 8.2 (2.4) | 8.1 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 5 | 8 | 20
  Male | 31 | 26 | 27 | 24 | 108
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 32 | 32 | 128

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Attention Deficit Hyperactivity Disorder (ADHD) Respondents
Description: Respondents were defined as having ≥30% decrease on the SNAP and CGI-I<=2). The Swanson, Nolan, and Pelham (SNAP)-IV Parent and Teacher Rating Scales were used to measure ADHD and oppositional symptoms at home and school. The SNAP-IV ADHD section contains items for each of the 18 Diagnostic and Statistical Manual of Mental Disorders-IV symptoms of ADHD rated from 0 (not at all) to 3 (very much). The Clinical Global Impressions Scale (CGI) includes subscales for severity of illness and global improvement. The Severity scale is scored from 1 (normal) to 7 (extremely ill), with a rating of ≥4 required for inclusion. The Improvement score ranged from 1 (very much improved) through 4 (no change) to 7 (very much worse). The CGI was completed by a blinded rater based on parent/child interview and review of completed parent and school behavior problem questionnaires at each study visit.
Time Frame: week 10
Measure: Number; unit: percentage of participants
Arm/Group | Atomoxetine + Parent Management Training | Atomoxetine Without Parent Management Training | Placebo + Parent Management Training | Placebo Without Parent Management Training
Number analyzed (Participants) | 32 | 32 | 32 | 32
percentage of participants | 45.2 | 46.9 | 29.0 | 19.4
Statistical Analysis 1: Comparison: Atomoxetine + Parent Management Training vs Atomoxetine Without Parent Management Training vs Placebo + Parent Management Training vs Placebo Without Parent Management Training; Test type: Superiority or Other; p = 0.47, Chi-squared

2. Primary Outcome: Percentage of Participants Who Were Autism Spectrum Disorder Respondents
Description: Respondents were defined as having ≥30% decrease on the HSQ and CGI-I≤2). The 25-item HSQ was adapted by the Research Units on Pediatric Psychopharmacology Autism Network to evaluate behavioral noncompliance in children with autism spectrum disorder (ASD). The Home Situations Questionnaire - Pervasive Developmental Disorder (HSQ) is a 25-item parent rating scale assessing noncompliance. Parents are asked to indicate whether each item is a problem and, if so, its severity from 1 (mild) to 9 (severe). The School Situations Questionnaire (SSQ) is a 9-item teacher rating scale that assesses noncompliance. The SSQ is a companion instrument to the HSQ and uses the same rating scale.
  The Clinical Global Impressions Scale (CGI) includes subscales for severity of illness and global improvement. The Severity scale is scored from 1 (normal) to 7 (extremely ill),
Time Frame: week 10
Measure: Number; unit: percentage of participants
Arm/Group | Atomoxetine + Parent Management Training | Atomoxetine Without Parent Management Training | Placebo + Parent Management Training | Placebo Without Parent Management Training
Number analyzed (Participants) | 32 | 32 | 32 | 32
percentage of participants | 22.6 | 43.8 | 38.7 | 16.4
Statistical Analysis 1: Comparison: Atomoxetine + Parent Management Training vs Atomoxetine Without Parent Management Training vs Placebo + Parent Management Training vs Placebo Without Parent Management Training; Test type: Superiority or Other; p = 0.95, Chi-squared

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: Only AEs related to study drug were assessed. Therefore AEs are presented for subjects on ATX or on placebo and not by arm. AEs were assessed for subjects taking at least one week of treatment. One participant in the ATX arm and two participants in the placebo arm did not take treatment for at least one week.
Groups:
- Atomoxetine: Data includes both the ATX alone arm and the ATX+ parent therapy arm
- Placebo: Data includes the placebo alone arm and the placebo+parent therapy arm
Arm/Group | Atomoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/62
Other Adverse Events (participants affected / at risk) | 59/63 | 61/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atomoxetine (N=63) | Placebo (N=62)
Irritability (Psychiatric disorders) | 27 | 29
Decreased Appetite (Metabolism and nutrition disorders) | 30 | 18
Agitation (Psychiatric disorders) | 19 | 20
Difficulty sleeping (General disorders) | 19 | 11
Vomiting (Gastrointestinal disorders) | 14 | 10
Constipation (Gastrointestinal disorders) | 7 | 9
Abdominal pain (Gastrointestinal disorders) | 10 | 3
Diarrhea (Gastrointestinal disorders) | 3 | 4
Aggression (Psychiatric disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No